CLINICAL TRIAL: NCT04955223
Title: Non-random Single-arm Clinical Study of Yinhu Qingwen Granule in the Treatment of Viral Pneumonia
Brief Title: Yinhu Qingwen Granule in the Treatment of Viral Pneumonia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHQWKL V2.0
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Viral Pneumonia
MeSH Terms: conditions — Pneumonia, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yinhu Qingwen Granule (Experimental): For mild and common patients, take 1 bag 2 times a day. For severe patients, take 1 bag 3 times a day. All treatment should be used for 10 days unless all the symtopms of patient with the viral pneumonia are relieved.
  Interventions: Drug: Yinhu Qingwen Granules

INTERVENTIONS:
Drug: Yinhu Qingwen Granules — For mild and common patients, take 1 bag 2 times a day. For severe patients, take 1 bag 3 times a day.

SUMMARY:
This is a non-randomized single arm clinical study to observe the effect of Yinhu Qingwen Granule in the relief of fever and improvement of related-symptoms of patients with viral pneumonia.

DETAILED DESCRIPTION:
Preliminary pharmacodynamic and toxicological studies can show that Yinhu Qingwen Granule has a certain effect on pneumonia caused by various viruses, and its safety is good. This study aims to observe the effect of Yinhu Qingwen Granule in the relief of fever and improvement of related-symptoms of patients with viral pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of viral pneumonia;
* Clinical diagnosis of Shi-du-yun-jie Zheng (damp stagnation syndrome) according to Chinese medicine, including fever,cough,sore throat,stuffy chest,irritability and thirst,short yellow urine,constipation or loose stool,thick and greasy yellow coating,and slippery pulse;
* Chest CT showed signs of acute exudative pneumonia in the lungs;
* Over 18 years old, regardless of gender, voluntarily signed an informed consent form;
* Those who were hospitalized and were accompanied by fever (body temperature ≥37.3℃) and respiratory tract symptoms like cough or dyspnea, when they were enrolled.

Exclusion Criteria:

* Patients that are susceptible to sensitivity or known to be allergic to the study drug;
* Patients whose white blood cell count ≥12×10^9 or neutrophil percentage ≥80%;
* Patients whose weight is less than 40 kg;
* Patients with respiratory failure or need mechanical ventilation;
* Patients with shock;
* Patients required to be in ICU monitoring and treatment;
* Patients participated in other clinical trials within 1 month;
* Patients with known renal impairment;
* Patients with any of the following laboratory parameter abnormalities during the screening period or within 24 hours before screening: ALT or AST level> 5 times the upper limit of normal range (ULN) or-ALT or AST level > 3 times ULN and total bilirubin level> 2 times ULN;
* Patients with immune system diseases and long-term use of immunosuppressive agents;
* Pregnant or breastfeeding women, or who have a positive pregnancy test during the screening period, or plan to become pregnant within 3 months after the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to the normalization of the temperature | up to 30 days
  The normalization of the temperature is defined as that the temperature of the patient dropped to normal and stabilized for more than 72 hours.

SECONDARY OUTCOMES:
Time to cough reported as mild or absent | Baseline, Day 3, Day 7, Day 10 and Day 30
  The severity of cough is assessed using Cough Symptom Scale, a scale range from 0-6. 0: cough absent;1-2: mild; 3-4:moderate; 5-6: severe
Mean clinical recovery time (hours) | up to 30 days
  The clinical recovery time is defined as the time from initiation of study treatment (active or placebo) until normalisation of fever, respiratory rate, and oxygen saturation, and alleviation of cough, sustained for at least 72 hours.
  Normalisation and alleviation criteria:
  (1) Fever: ≤36.6°C or -axilla, ≤37.2 °C oral or ≤37.8°C rectal or tympanic;(2)Respiratory rate - ≤24/minute on room air; 3) Oxygen saturation - >94% on room air; (4) Cough - mild or absent on a patient reported scale (cough symptoms score ≤ 2 points).
Time to dyspnea reported as mild or absent | Baseline, Day 3, Day 7, Day 10 and Day 30
  The severity of dyspnea is assessed on a self-reported scale of severe, moderate, mild or absent.
Mean blood oxygen saturation | Baseline, Day 3, Day 7, Day 10
Mean neutrophil/lymphocyte ratio (NLR) | Baseline, Day 10
  Neutrophil/lymphocyte ratio (NLR) is obtained from the blood routine.
Frequency of requirement for supplemental oxygen or non-invasive ventilation | up to 30 days
Mean time of supplemental oxygen (days) | up to 30 days
Mean time of non-invasive ventilation (days) | up to 30 days
Severe case incidence | up to 30 days
  Severe case is defined as respiratory rate ≥30/minute on room air；or Oxygen saturation - ≤94% on room air；or PaO2/FiO2≤300mmHg.
Proportion of re-hospitalization or admission to ICU | up to 30 days
All-cause mortality | up to 30 days
Frequency of serious adverse events | up to 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Chengdu First People's Hospital/Chengdu integrated TCM & Western Medicine Hospital, Chengdu, Sichuan